CLINICAL TRIAL: NCT06370611
Title: Early REmote Rehabilitation to Improve Health of the Elderly After CARDiac Surgery. (RECARD Trial). A Bi-center, Prospective, Randomized, Open-label, Blinded Evaluation (PROBE) Trial
Brief Title: Early Remote Rehabilitation to Improve Health of the Elderly After Cardiac Surgery. (RECARD Trial)
Acronym: RECARD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ivy susanne Modrau, MD (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Sponsor-Investigator, Ivy susanne Modrau, MD, Dr. Med., Consultant Cardiac Surgon, Associate Professor, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2314027
Record Dates: First submitted 2024-04-08; First posted 2024-04-17 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Cardiac Rehabilitation
Keywords: Cardiac Surgery; Mobile Health; Elderly; Exercise; Randomised Controlled Trial
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Bi-center, prospective, randomized, controlled, parallel (1:1), two-arm, open-label, blinded evaluation (PROBE) trial
Who Masked: Outcomes Assessor
Masking Description: Allocation cannot be concealed from the participants, care providers or investigator. Outcome assessors will be blinded regarding allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early mobile health intervention (Active Comparator): ICURA app and sensor-based technology, individualized training plan, and weekly calls from a physiotherapist in addition to standard care
  Interventions: Device: Early mobile health intervention supplemented by weekly calls from a physiotherapist
- Control (No Intervention): Standard care consists of physiotherapy group education of about 10-15 minutes regarding mobilization, respiratory therapy, and sternal precautions after surgery. After surgery, phase I in-hospital rehabilitation consists of respiratory therapy, mobilization from supine and sitting position, and walking down a corridor. Prior to discharge, all patients are encouraged to undertake daily walks and resume activities of daily living, and engage in recommended moderate physical activity (Borg's scale 12-14). All patients are referred to CR in their municipality.

INTERVENTIONS:
Device: Early mobile health intervention supplemented by weekly calls from a physiotherapist — Six-week home-based rehabilitation program using the ICURA app and sensor-based technology (ICURA ApS, Copenhagen, Denmark). During the hospital stay patients in the intervention group are introduced to the app's usage, and an individualized training plan is collaboratively created and subsequently tailored by a physiotherapist.
  The comprehensive mobile health intervention includes customized training programs, activity tracking, visualization of exercises with videos, and a password-protected webpage for physiotherapists to customize training programs and track patient activity.
  The patients will receive two calls from a physiotherapist per week for the first two weeks and as required the following four weeks.
  Other Names: ICURA
  Arms: Early mobile health intervention

SUMMARY:
An increasing number of older patients undergo heart surgery. Despite seemingly successful outcomes, these vulnerable patients may face prolonged decreased functional capacity, reduced self-efficacy, and impaired quality of life after discharge. Early engagement in physical activity and education plays a key role in health and well-being after heart surgery The goal of this clinical trial is to evaluate the effectiveness of an app-based exercise program and weekly calls from a physiotherapist in the early stages after open heart surgery.

Eligible patients will be randomly assigned to either a control group receiving standard care or an intervention group, which will be introduced to an individually tailored exercise program as an addition to standard care.

Follow-up is planned with an out-patient visit six weeks after discharge and a telephone interview six months post-surgery.

All participants will undergo assessments at enrollment and during follow-up. Physical performance will be evaluated through physical tests. General well-being, quality of life, self-reported physical activity, and cost-effectiveness of the intervention will be assessed through questionnaires. Muscle health will be examined through blood sampling, CT scans, and muscle biopsies.

The primary endpoint is the 30-second Chair Stand Test serving as a measurement of physical function.

DETAILED DESCRIPTION:
Hypotheses:

Primary: Early mobile health intervention at home supplemented by weekly calls from a physiotherapist after cardiac surgery improves functional outcomes, exercise tolerance, and quality of life in older patients.

Secondary:

* Cardiac surgery increases the prevalence and extent of sarcopenia in the elderly which can be mitigated by early mobile health intervention
* Sarcopenia on Chest Computed Tomography (CCT) is strongly correlated to functional outcome and quality of life following cardiac surgery
* Early mobile health intervention is feasible and cost-effective

Design:

This is a bi-center, prospective, randomized controlled, parallel, two-arm, open-label, blinded evaluation (PROBE) trial with a superiority design. The study population will consist of a representative group (n=120) of older patients scheduled for open heart surgery who fulfill the requirements according to inclusion and exclusion criteria. The patients will be recruited from 2 cardiac surgery centers in northern and central Denmark.

Patients are stratified after center and subsequently randomly allocated (1:1) to receive mobile health intervention as an adjunct to standard care (Intervention Group), or standard care alone (Control group) for 6 weeks after discharge. Follow-up is planned with an outpatient visit 6 weeks after discharge, and a telephone interview 6 months after surgery.

Patients in the intervention group receive a 6-week home-based CR using the ICURA app and sensor-based technology (ICURA ApS, Copenhagen, Denmark). During the hospital stay patients in the intervention group are introduced to the app's usage, and an individualized training plan is collaboratively created and subsequently tailored by a physiotherapist. The patients are equipped with a case including an ICURA -sensor with a charger, an illustrative quick guide, and a contact telephone number. According to the patient's preference, the app is either installed on their own mobile phone or provided on a separate mobile device.

The comprehensive mobile health intervention includes customized training programs, activity tracking, visualization of exercises with videos, text message communication with patients, and a password-protected webpage for physiotherapists to customize training programs and track patient activity.

A few days after discharge, patients in the intervention group will receive the first call from the physiotherapist, to ensure, that the patient is using the ICURA app actively. The patients will receive two calls per week for the first two weeks and as required the following four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Scheduled first-time heart surgery through median sternotomy
* Male or female, aged ≥ 65 years (The age criterion implies the exclusion of women of childbearing potential)

Exclusion Criteria:

* Medical conditions requiring referral to specialized rehabilitation (e.g., severe heart or lung failure, need for blood pressure monitoring during exercise)
* Emergent procedure
* Anticipated inability to perform intervention, study assessment procedures, or follow-up
* Participation in any other interventional clinical that may interfere with the outcome measures

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change (Δ) 30-second chair stand test (30CST) baseline vs. 6-week FU | 1-7 days prior to surgery and 6 weeks (+/- 4 days) after surgery
  Recording of the number of stands a person can complete from a chair without arms in 30 seconds

SECONDARY OUTCOMES:
Change (Δ) in 10-meter Walk Test (10MWT) baseline vs. 6-week FU | 1-7 days prior to surgery and 6 weeks (+/- 4 days) after discharge
  Measurement of walking speed in meters per second over a 10-meter distance
Difference in 6-minute Walk Test (6MWT) between groups at 6-week FU | 6 weeks (+/- 4 days) after discharge
  Measurement of walking distance in 6 minutes.
Change (Δ) in WHO-5-score baseline vs. 6-week FU | 1-7 days prior to surgery and 6 weeks (+/- 4 days) after discharge and 6 months after surgery
  5-item World Health Organization Well-Being Index (WHO-5), questionnaire assessing subjective well-being
Change (Δ) in ASS-2-score baseline vs. 6-week FU | 1-7 days prior to surgery and 6 weeks (+/- 4 days) after discharge and 6 months after surgery
  Anxiety Symptom Scale-2 (ASS-2), questionnaire assessing anxiety
Change (Δ) in MDI-2-score baseline vs. 6-week FU | 1-7 days prior to surgery and 6 weeks (+/- 4 days) after discharge and 6 months after surgery
  Major Depression Inventory-2 (MDI-2), questionnaire assessing depression
Change (Δ) in Self-reported Physical Activity baseline vs. 6-week FU | 1-7 days prior to surgery and 6 weeks (+/- 4 days) after discharge and 6 months after surgery
  Questionnaire assessing self-reported physical activity
Change (Δ) in EuroQol-score baseline vs. 6-week FU | 1-7 days prior to surgery and 6 weeks (+/- 4 days) after discharge and 6 months after surgery
  EuroQol-5-Dimension-5-Level Questionnaire (EQ-5D-5L), questionnaire assessing health-related quality of life
Change in skeletal muscle mass baseline vs. 6-week FU | 1-7 days prior to surgery and 6 weeks (+/- 4 days) after discharge
  Body composition analysis with artificial-intelligence-assisted medical image analysis (CT scan) (DAFS©, Veronoi Health Analytics, Vancouver, Canada) to assess quantity and quality of skeletal muscle.
Cost-effectiveness analysis | 1-7 days prior to surgery and 6 weeks (+/- 4 days) after discharge and 6 months after surgery
  Questionnaire assessing the cost-effectiveness of the intervention in comparison to usual care
Changes in markers of musculoskeletal health through blood samples baseline vs. 6-week FU | 1-7 days prior to surgery and 6 weeks (+/- 4 days) after discharge
  Markers of muscle health: Myoglobin, Creatine Kinase (CK)
Changes in markers of inflammation through blood samples baseline vs. 6-week FU | 1-7 days prior to surgery and 6 weeks (+/- 4 days) after discharge
  Inflammatory markers: White Cell Count (WCC), Platelet Count, Mean Platelet Volume (MPV), Immature Platelet Fraction (IPF), High-Sensitive C-Reactive Protein (hs-CRP)
Changes in markers of nutrition through blood samples baseline vs. 6-week FU | 1-7 days prior to surgery and 6 weeks (+/- 4 days) after discharge
  Nutritional markers: Hemoglobin, Glycated Hemoglobin (HbA1c), fasting glucose, Albumin, Triglycerides, High-Density Lipoprotein (HDL), Low-Density Lipoprotein (LDL), Vitamin B12, Folate, 25-OH-Vitamin D2+D3
Changes in markers of liver function through blood samples baseline vs. 6-week FU | 1-7 days prior to surgery and 6 weeks (+/- 4 days) after discharge
  Liver Function Markers: Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT)
Changes in markers of kidney function through blood samples baseline vs. 6-week FU | 1-7 days prior to surgery and 6 weeks (+/- 4 days) after discharge
  Kidney Function Markers: Creatinine, estimated Glomerular Filtration Rate (eGFR)
Changes in markers of hormone levels through blood samples baseline vs. 6-week FU | 1-7 days prior to surgery and 6 weeks (+/- 4 days) after discharge
  Hormonal Markers: Cortisol, Free/Total Testosterone, Sex Hormone Binding Globulin (SHBG), Insulin-like Growth Factor-1 (IGF-1)
Assessment of muscle quality through obtainment of biopsies of the pectoralis major muscle at the surgery | At surgery
  Analysis of pectoralis major muscle biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Ivy S. Modrau, MD, dr.med., Study Chair — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aarlborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus

IPD SHARING:
Plan to Share IPD: No
The participants of this study did not give written consent for their data to be shared publicly, so due to the sensitive nature of the research supporting data is not available.

REFERENCES:
- [Derived] Daugaard R, Sorensen L, Ingemann-Molden S, Modrau IS. Early remote rehabilitation to improve health of the elderly after cardiac surgery - study protocol for a randomised trial. Dan Med J. 2025 Jun 21;72(7):A11240820. doi: 10.61409/A11240820. PMID 40600679